CLINICAL TRIAL: NCT01038154
Title: Randomized Controlled Study to Evaluate the Efficacy of Pravastatin on Survival and Recurrence of Advanced Gastroesophageal Cancer
Brief Title: Study to Evaluate the Efficacy of Pravastatin on Survival and Recurrence of Advanced Gastroesophageal Cancer
Acronym: AGIM-1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Donostia (Other)
Responsible Party: Luis Bujanda. Department of Gastroenterology. Hospital Donostia. Osakidetza., Luis Bujanda. Department of Gastroenterology. Hospital Donostia. Osakidetza.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AGIM-1
Record Dates: First submitted 2009-12-02; First posted 2009-12-23 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2009-12

CONDITIONS: Esophageal Cancer; Stomach Cancer
Keywords: advanced esophageal cancer and stomach cancer; Pravastatin; Survival; adverse effects
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms | interventions — Pravastatin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): Not Receive pravastatin
- Pravastatin (Experimental)
  Interventions: Drug: Pravastatin

INTERVENTIONS:
Drug: Pravastatin — Receive one tablet of 40 mg of pravastatin, orally every 24 hours (at breakfast) for 2 years.
  Other Names: esophageal cancer and stomach cancer
  Arms: Pravastatin

SUMMARY:
The survival of esophageal cancer and stomach cancer (EGC) at 5 years is less than 30%. Pravastatin is a potent inhibitor of HMG-CoA reductase inhibitor that has shown increased survival in patients with advanced hepatocellular carcinoma. The objective is to evaluate the efficacy of treatment (increase in survival and recurrence-free period of the disease) with pravastatin in patients with advanced EGC. The investigators have designed a randomized, controlled and open. Advanced stage was considered for patients with T4 or N1 or M1 according to the TNM classification. It has been estimated sample size per treatment arm of 73 patients (146 patients in total). Randomization was done on a stratified by location (CE or CG). All patients receive hatitual treatment (surgery and / or chemotherapy and / or radiotherapy and / or palliative) for each of their clinical conditions. The experimental group will receive one tablet of 40 mg of pravastatin orally every 24 hours (breakfast) for 2 years. There will be a monthly monitoring of these patients for at least 2 years which includes an analytics. Every 2 months there will be an abdominal-pelvic CT scan to assess progression and treatment response.

DETAILED DESCRIPTION:
1. Design: A randomized, controlled, open, parallel group study to assess the survival and disease-free period or progression in patients with advanced CGE over a period of 2 years.
2. Under study: Patients diagnosed in histology for the first time, advanced-stage CGE and fulfilling the inclusion criteria and none of the exclusion criteria proposed in the Hospital Donostia (San Sebastian) and Hospital de Basurto (Bilbao) .
3. Inclusion criteria: older than 18 years, esophageal or gastric cancer histologically confirmed (squamous or adenocarcinoma) for the first time, advanced stage (T4 or N1 or M1) according to the fourth edition of TNM classification and signing the informed consent
4. Exclusion criteria: Patients who routinely take (more than 3 days a week) anti-inflammatory drugs or aspirin, patients receiving oral anticoagulants, fibrates, cyclosporine and oral contraceptives, patients with hypersensitivity to pravastatin, pregnant women being lactation, peripheral neuropathy grade 2 or greater, patients who have been diagnosed in the previous 5 years other than skin cancer tumor that is not melanoma or carcinoma in situ of cervix or bladder, patients receiving chemotherapy or radiotherapy for other of tumor patients in their laboratory parameters before starting the present study transaminases or alkaline phosphatase more than twice the normal value, patients with platelet count less than 100.000/mm3, absolute neutrophil count below 1000/mm3, or patients with evidence of bleeding diathesis or coagulopathy, patients with heart failure than NYHA grade II, patients with creatinine greater than 2 mg / dL, patients over 75 years, asthmatics, patients with physical or mental disability, patients with alcoholism or patients with diseases hereditary muscle
5. Intervention: Patients were randomized to two groups:

   * Experimental Group: You will receive one tablet of 40 mg of pravastatin Cinfa EFG, orally every 24 hours (at breakfast) for 2 years.
   * Control Group: will not receive pravastatin. All patients receive the prescribed treatment (surgery and / or chemotherapy and / or radiotherapy and / or palliative) based on their stage and clinical situation.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years,
* Esophageal or gastric cancer histologically confirmed (squamous or adenocarcinoma) for the first time,
* Advanced stage (T4 or N1 or M1) according to the fourth edition of TNM classification,
* Signing the informed consent.

Exclusion Criteria:

* Patients who routinely take (more than 3 days a week) anti-inflammatory drugs or aspirin,
* Patients receiving oral anticoagulants, fibrates, cyclosporine and oral contraceptives,
* Patients with hypersensitivity to pravastatin,
* Pregnant or lactating women,
* Peripheral neuropathy grade 2 or greater,
* Patients who have been diagnosed in the previous 5 years other than skin cancer tumor that is not melanoma or carcinoma in situ of cervix or bladder,
* Patients receiving chemotherapy or radiotherapy for another type of tumor,
* Patients in their laboratory parameters before starting the present study transaminases or alkaline phosphatase more than twice the normal value,
* Patients with platelet count less than 100.000/mm3, absolute neutrophil count below 1000/mm3,
* Patients with evidence of bleeding diathesis or coagulopathy,
* Patients with heart failure than NYHA grade II,
* Patients with creatinine greater than 2 mg / dL,
* Patients over 75 years,
* Asthmatics,
* Patients with physical or mental disability,
* Patients with alcoholism, OR
* Patients with hereditary muscle disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
all cause mortality | two years

SECONDARY OUTCOMES:
free time of disease recurrence | two years

CONTACTS AND LOCATIONS:
Overall Officials: Luis Bujanda, Prof., Principal Investigator — Osakidetza
Locations (1):
- Department Gastroenterology. Hospital Donostia, San Sebastián, Guipúzcoa, Spain